CLINICAL TRIAL: NCT07014956
Title: Intelligence and Neurodevelopmental Outcome After Prenatal Exposure to Labour Epidural Analgesia: a Sibling Matched Clinical Ambidirectional Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S69530
Record Dates: First submitted 2025-05-19; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Pregnancy; Epidural Analgesia, Obstetric
Keywords: Labour epidural analgesia; Neurodevelopmental outcome; Intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed: Children prenatally exposed to labour epidural analgesia
  Interventions: Procedure: Labour epidural analgesia
- Unexposed: Prenatally not exposed to labour epidural analgesia

INTERVENTIONS:
Procedure: Labour epidural analgesia — Prenatal exposure to labour epidural analgesia during delivery
  Groups: Exposed

SUMMARY:
In Belgium, labour epidural analgesia (LEA) has been used for decades in the vast majority of vaginal deliveries (up to 83% of deliveries). Labour epidural analgesia is the most effective and safest way to allow pregnant women a nearly pain-free labour- and birth experience. Recent data showed that the use of LEA was associated with a reduced risk for severe maternal morbidity, neonatal resuscitation and with a reduced risk for low Apgar scores. However, prenatal exposure to labour epidural analgesia has been associated by several study groups with an increased risk for autism spectrum disorder (ASD) in the children, but these studies suffer from several important limitations which may have induced significant bias (e.g., not correcting for unmeasured confounders). Associations with other neurodevelopmental disorders (e.g., Attention Deficit Hyperactivity Disorder (ADHD), oppositional defiant disorder (ODD) and conduct disorder (CD)) and cognitive functioning have not been investigated yet. There is hence an urgent need for a study allowing definitive conclusions by overcoming the limitations of the previous studies. The investigators will perform the first sibling-matched clinical cohort study using a prospective investigator-assessment of multiple domains of cognitive functions. The investigators hypothesize that prenatal exposure to LEA will neither be associated with reduced intelligence nor with more neurodevelopmental disorders. Validating this hypothesis holds the potential to grant women the assurance to confidently receive the most efficacious method for labour analgesia, free from apprehension that it might have adverse implications for their children's neurodevelopment.

DETAILED DESCRIPTION:
Primary objective:

To compare the intelligence of children prenatally exposed to labour epidural analgesia with that of sibling matched unexposed children.

Secondary objective(s):

To compare parentally reported traits of ASD, ADHD, ODD and CD of children prenatally exposed to labour epidural analgesia with that of sibling matched unexposed children.

Endpoints:

* Primary endpoint: Wechsler full scale intelligence quotient
* Secondary endpoints: multiple indexes assessed by the Wechsler intelligence scale: verbal comprehension index, visual spatial index, working memory index, fluid reasoning index and processing speed index. Total scores and subscores of the parental questionnaires "social responsiveness scale" (SRS) and "vragenlijst voor gedragsproblemen bij kinderen 6-16" (VvGK6-16) are additional secondary endpoints.

Sample size:

At least 64 prenatally exposed children and 64 prenatally unexposed children

Summary of eligibility criteria:

Dutch speaking sibling pairs discordant for prenatal exposure to labour epidural analgesia will be included. Children born from 1st January 2014 until 1st November 2019 will be included. Children prenatally exposed to maternal surgery, foetal surgery/interventions, chemotherapy, radiotherapy, radiology and oncologic pathology will be excluded. Children with a diagnosis of severe disability of genetic origin (e.g., Fragil X, Down syndrome,…), history of head trauma, major congenital birth defects, children born at a gestational age < 37 weeks or > 42 weeks, or with a birth weight < 2.5 kg will be excluded. Children exposed to general anaesthesia after birth, twins/triplets/multiple births will be excluded. Elective and intrapartum caesarean sections will be excluded.

Maximum duration a research subject remains in the study:

Study will be conducted in 2024-2027. The end of the study for each individual participant is determined by the date at which the neuropsychological testing is planned. Neuropsychological testing usually takes no longer than 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Exposed children: Children prenatally exposed to labour epidural analgesia
* Unexposed children: Sibling of an exposed child, Prenatally not exposed to labour epidural analgesia
* Exposed & unexposed children: Children born from 1st January 2014 until 1st November 2019, Parental informed consent

Exclusion Criteria:

* Children whose mothers underwent maternal surgery or foetal surgery/interventions during the same pregnancy.
* Children exposed to general anaesthesia after birth
* Children prenatally exposed to chemotherapy, radiotherapy, radiology, oncologic pathology
* Children born at a gestational age < 37 weeks or > 42 weeks, or with a birth weight < 2.5 kg
* Twins, triplets, multiple births
* No Dutch-speaking children
* Diagnosis of severe disability of genetic origin (e.g., Fragil X, Down syndrome,…), history of head trauma, major congenital birth defects
* Elective caesarean section and intrapartum caesarean section (the number of caesarean sections will be reported and compared between both groups)
* Foetus died before start of delivery

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Sibling pairs discordant for prenatal exposure to labour epidural analgesia will be included
Sampling Method: Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Wechsler full-scale intelligence quotient | At te moment of neuropsychological testing
  Will be assessed using the Wechsler Intelligence Scale for Children (WISC). Minimum value: 40, maximum value: 160. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Indices of the Wechsler intelligence scale | At te moment of neuropsychological testing
  Verbal comprehension, working memory, visual spatial, fluid reasoning, processing speed. Minimum value: 40, maximum value: 160. Higher scores mean a better outcome.
Clinically relevantly decreased intelligence quotient | At te moment of neuropsychological testing
  The absolute risk reduction for a clinically relevantly decreased intelligence quotient, defined as an IQ<85, will be calculated.
Social responsiveness scale (SRS) | At te moment of neuropsychological testing
  Parental reported social deficits in the autism spectrum. Minimum value: 0, maximum value: 195. Higher scores represent a worse outcome.
Disruptive Behavior Disorders Rating Scale (DBDRS) | At te moment of neuropsychological testing
  Parental reported traits of inattention, hyperactivity and impulsivity (ADHD), oppositional defiant disorder (ODD) and conduct disorder (CD). Minimum value: 0, maximum value: 135. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Can be requested from authors.
Supporting Information: Study Protocol
Time Frame: Can be requested from authors.
Access Criteria: Can be requested from authors.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT07014956/Prot_SAP_000.pdf